CLINICAL TRIAL: NCT01744834
Title: Learning in Young Adults as Predictor for the Development of Alcohol Use Disorders
Acronym: LeAD
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: HE2597/13-1;SM80/71;WI709/10-1
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: High-risk Alcohol Consumption Pattern; Low-risk Alcohol Consumption Pattern
Keywords: Reward-based learning; Pavlovian-to-instrumental transfer; Functional imaging; alcohol use disorder risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsample are taken for genetic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 18-year-old males: 18-year-old males, representative random sample of the Dresden/Berlin (Germany) area, categorized as high and as low-risk drinkers respectively

SUMMARY:
Overall goal of this study is to scrutinize the relation of learning behavior and related brain activity to the development of alcohol use disorder (AUD).

The researchers aim is to characterise a representative sample (200 men at age 18) with regard to learning parameters and their respective neural correlates which are thought to be indicators for the risk to develop an alcohol use disorder.

As part of a large multi-center study on alcohol dependency (in Dresden & Berlin, Germany) the researchers will characterize the sample and then prospectively assess alcohol consumption and development of AUDs over a period of three years plus additional follow-ups after that period, depending on future funding.

Among other hypotheses it is expected that increased activation of striatal and prefrontal brain regions by the Pavlovian-to-instrumental transfer process is related to increased risk of developing an AUD.

DETAILED DESCRIPTION:
Hazardous alcohol use and alcohol use disorders (AUDs) are extremely prevalent in industrialized countries, affecting about 6 million individuals in Germany alone. The onset of most cases occurs during adolescence and early adulthood. Therefore, targeted prevention would be desirable especially in young people who are at high risk to develop AUDs. Since our knowledge about predisposing factors is limited, this project aims to identify mechanisms underlying liability for dysfunctional alcohol consumption (i.e. hazardous alcohol use, alcohol abuse and alcohol dependence). Based on the hypothesis that addiction is a disorder due to aberrant learning, the researchers expect that inter-individual differences in learning behavior should be associated with liability for as well as resiliency against AUD. To test the hypotheses, the researchers will characterize 200 men at age 18, and then prospectively assess alcohol consumption and development of AUDs over a period of three years. At baseline, the researchers will study three clusters of predictive variables: (i) individual learning parameters, estimated by computational modeling of behavioral performance in learning tasks such as Pavlovian-to-instrumental transfer, probabilistic reversal learning, and habitization-devaluation; (ii) individual neural correlates of learning, assessed by functional brain imaging during learning; and (iii) already established risk factors such as family history of alcoholism and impulsivity.

The specific aim is to test a set of related hypotheses. The researchers assume that high risk for AUD at baseline (cross-sectional design), increase of alcohol consumption after 3 years and incidence or progression of AUD during follow-up (prospective data) will be associated with decreased reward sensitivity, decreased punishment sensitivity, increased Pavlovian approach behavior ('sign tracking'), increased 'go' effect of conditioned appetitive stimuli, increased habitization, increased activation of striatal and prefrontal brain regions by the Pavlovian-to-instrumental transfer process, decreased correlation between striatal brain activity and prediction error during reversal learning.

ELIGIBILITY:
Inclusion Criteria:

* men at age 18
* ability to provide fully informed consent and to use self-rating scales
* habitual social drinking during the three months preceding participation, defined by at least two drinking days in any four weeks-interval
* being able to provide information concerning biological parents and grandparents

Exclusion Criteria:

* lifetime history of Diagnostic Statistical Manual-IV bipolar or psychotic disorder
* current diagnosis of one of the following disorders: major depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder, or obsessive-compulsive disorder
* prior treatment for any axis-I or axis-II disorder except for specific disorders of childhood and adolescence (i.e., oppositional defiant disorder, conduct disorder, ADHD)
* history of substance dependence other than nicotine dependence
* current substance use other than nicotine and alcohol as evinced by positive urine screen
* history of severe head trauma or other severe central neurological disorder (e.g. multiple sclerosis)
* any alcohol intake in the last 24 hours before test days
* use of medications or illicit substances known to interact with the central nervous system within the last 10 days or at least four half-lives post last intake

Ages: 18 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: random, representative sample from the respective city area (100 in Dresden, 100 in Berlin; male; born between January 1 1994 and November 30 1994
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2012-12; Primary Completion 2018-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
blood oxygenation level dependent (BOLD) response | time point 1: when subject is 18 years of age
  investigation of neural activation of the mesolimbic system in a healthy random sample of male subjects categorized in high and low risk-for-AUD using 3 Tesla magnetic resonance imaging

SECONDARY OUTCOMES:
alcohol consumption pattern after and during a 3-year follow-up period | assessment every 6 months
  time life follow-back assessment of alcohol consumption pattern will be assessed every 6 months, as well as standardized diagnostic interviewing for psychopathologies every 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smolka, Prof MD, Principal Investigator — Technische Universität Dresden, Dresden, Germany; Andreas Heinz, Prof MD, Principal Investigator — Charité University, Berlin, Germany; Andreas Heinz, Prof MD, Study Chair — Charité University, Berlin, Germany; Hans-Ulrich Wittchen, Prof PhD, Study Director — Technische Universität Dresden, Dresden, Germany
Locations (3):
- Germany (3):
  - Technische Universität Dresden, Dresden, Saxony
  - Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin

REFERENCES:
- See also: English study description — http://gepris.dfg.de/gepris/projekt/209288318